CLINICAL TRIAL: NCT06608238
Title: A Randomized, Double-Blinded, Placebo Controlled Trial to Evaluate the Safety and Efficacy of a Doxorubicin Microneedle Array (D-MNA) for the Treatment of Nodular Basal Cell Carcinoma in Adults
Brief Title: The Purpose of This Study is to Evaluate the Safety and Efficacy of D-MNA in Adult Patients With Nodular Basal Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SkinJect, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SKNJCT-003
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Nodular Basal Cell Carcinoma

STUDY DESIGN:
Intervention Model Description: 60 subjects randomized in a 1:1:1 ratio to receive placebo or one of the D-MNA doses weekly for three doses.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded (Participant and Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Active Comparator): D-MNA 200 mcg, intradermal patch, given once weekly for 2 weeks.
  Interventions: Drug: D-MNA 200 mcg
- Arm B (Active Comparator): D-MNA 100 mcg intradermal patch, given once weekly for 2 weeks
  Interventions: Drug: D-MNA 100 mcg
- Arm C (Placebo Comparator): P-MNA, intradermal patch, given once weekly for 2 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: D-MNA 200 mcg — D-MNA , (doxorubicin) patch, 200 mcg
  Arms: Arm A
Drug: D-MNA 100 mcg — D-MNA (doxorubicin) patch, 100 mcg
  Arms: Arm B
Other: Placebo — P-MNA patch, placebo
  Arms: Arm C

SUMMARY:
The goal of the study is to learn about the safety and how effective two different strengths of D-MNA compared to a placebo (a look-alike substance that contains no drug) in the treatment of nodular basal cell skin cancer

DETAILED DESCRIPTION:
A double-blind, randomized, placebo-controlled study designed to evaluate the safety and efficacy of D-MNA which is administered as an intradermal injection in subjects with nodular Basal Cell Carcinoma (nBCC).

About 60 subjects will be enrolled. Enrolled subjects will be randomly allocated to receive D-MNA or placebo injection on the identified target lesion once weekly for 3 weeks.

After two weeks, the target lesion will be excised.

An Interim Analysis will be done after 26-30 subjects would have completed Visit 5/ Excision Visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female ≥ 18 years of age.
2. Clinical diagnosis of a primary, previously untreated, histologically confirmed nodular Basal Cell Carcinoma (nBCC) lesion suitable for excision (at end of the study) with a minimum diameter of 0.5 cm and with a maximum longest diameter of 1.3 cm at the time of biopsy and Visit 2/Baseline.
3. Willing to refrain from exposure to excessive direct sunlight or ultraviolet light and to avoid the use of tanning beds for the duration of the study.
4. Willing and able to receive the test article treatments, comply with study instructions, and commit to all follow-up visits for the duration of the study.

Exclusion Criteria:

1. Pregnant, lactating, or planning to become pregnant.
2. nBCC is located on the face, scalp, digits, mucosa, or skin that is scarred or previously treated with radiation.
3. History of treated nBCC lesion recurrence or basal cell nevus syndrome.
4. Immunocompromised, based on medical condition (e.g., human immunodeficiency virus), medication use, or other factors.
5. Active malignancy, excluding non-metastatic prostate cancer, other cutaneous basal or squamous cell carcinomas, and carcinoma of the cervix.
6. Used systemic chemotherapeutic agents within the 12 months prior to Visit 2/Baseline.
7. Clinical laboratory results at Visit 1/Screening within the following ranges: (a) granulocytes < 2,000/mm3, (b) platelets <50,000/mm3, (c) serum creatinine greater than 2 times the upper limit of normal (ULN), (d) aspartate aminotransferase, alkaline aminotransferase, lactate dehydrogenase, or alkaline phosphatase greater than 3 times the ULN.
8. History of sensitivity to any of the ingredients in the test articles .

12. Used topical immunomodulators within 2 cm of the Target Lesion within the 4 weeks prior to Visit 2/Baseline or after the confirmatory biopsy.

9. Used the following topical agents within 2 cm of the Target Lesion within the 4 weeks prior to Visit 2/Baseline or after the confirmatory biopsy: aminolevulinic acid, 5-fluorouracil, diclofenac, ingenol mebutate, tirbanibulin, or imiquimod.

10. Has been treated with liquid nitrogen, surgical excision or curettage within 2 cm of the Target Lesion within 4 weeks prior to Visit 2/Baseline or after the confirmatory biopsy.

11. Currently enrolled in an investigational drug, biologic, or device study. 12. Used an investigational drug, investigational biologic, or investigational device treatment within 30 days prior to enrollment into the study.

13. Unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-02-05 (Estimated); Study Completion 2025-06-02 (Estimated)

PRIMARY OUTCOMES:
Histological Clearance of Target Lesion | 29 to 34 days from enrollment into the study
  Proportion of subjects with complete histological clearance of the Target Lesion at Visit 5/EV

SECONDARY OUTCOMES:
Clinical Clearance of Target Lesion | 29 to 34 days from enrollment into the study
  Proportion of subjects with complete clinical clearance of the Target Lesion at Visit 5/EV.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Site #4, Fresno, California
  - Site #6, San Diego, California
  - Site #1, Rolling Meadows, Illinois
  - Site #5, Mandeville, Louisiana
  - Site #3, Highlands, New Jersey
  - Site#2, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided